CLINICAL TRIAL: NCT04473118
Title: Burnout, Anxiety, Depression, Stress (BADS) and Post-Trauma Stress Disorder (PTSD) in Healthcare Workers Exposed to COVID-19 Patients
Brief Title: Assessment of Mental Health in Healthcare Workers Exposed to COVID-19 Patients
Acronym: BADS-PTSD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Ali Ait Hssain, Senior consultant intensivist, Hamad Medical Corporation
Other Study IDs: MRC-05-017
Record Dates: First submitted 2020-07-15; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: Mental health; Burnout; Anxiety; Depression; Stress; Post-trauma stress disorder; Healthcare workers
MeSH Terms: conditions — COVID-19; Psychological Well-Being; Burnout, Psychological; Anxiety Disorders; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare workers: All healthcare workers exposed directly or not to suspected or infected COVID-19 patients such as nurse; paramedic; senior physician; resident/ trainee physician; respiratory therapist; perfusionist; physiotherapist; dietitian; technician lab; technician imaging; pharmacist; occupational therapist; speech therapist
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — An online-based questionnaire sent to participants via email

SUMMARY:
The recent COVID-19 outbreak has put the health care workers on the frontline to interact and provide support to the patients. Based on previous disease outbreak-associated studies, it is evident that these individuals are at a high-risk of developing psychological distress such as burnout, anxiety, depression, and stress (BADS). Thus, the current study aims to evaluate the mental health outcomes of healthcare workers dealing with COVID-19 patients within Qatar and internationally, during and after the COVID-19 crisis. The participants will be divided into two groups: those working with COVID-19 patients and those not working with COVID-19 patients. The magnitude of symptoms of BADS will be assessed using electronic versions of the standardized questionnaires: Maslach Burnout Inventory (MBI-HSS), Hospital Anxiety and Depression Scale (HADS), Depression, Anxiety and Stress Scale (DASS-21), and Conditions for Work Effectiveness (CWEQ). A follow-up survey will be sent to both groups after the COVID-19 crisis to assess their vulnerability to develop post-trauma stress disorder (PTSD) using a PDS-5 survey.

DETAILED DESCRIPTION:
Coronaviruses belong to a large family of viruses, responsible for causing mild respiratory infections such as the common cold or severe syndromes such as the Middle East Respiratory Syndrome (MERS) or Severe Acute Respiratory Syndrome (SARS). A novel coronavirus named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is responsible for the most recent disease outbreak called COVID-19 that originated in Wuhan, China in December 2019. The outbreak rapidly spread to other parts of China and the world, including Qatar. As of 4th March 2020, the total number of confirmed cases in Qatar is 1325 and worldwide is 1,169,262. On 11 March 2020, the World Health Organization had declared COVID-19 as a global pandemic.

The health care workers are on the frontline providing routine and essential services to the COVID-19 patients, including diagnosis, treatment, and care. Consequently, these individuals are at a high risk of developing and experiencing psychological distress. Considering the continuously increasing suspected and confirmed COVID-19 cases, lack of specific treatment, inadequate personal protective equipment and the need for meticulous nursing care, the health care workers are overburdened mentally and are prone to mental illnesses. Not to mention, the risk of themselves getting infected due to direct exposure to patients and subsequent self-isolation they must undertake to prevent the spread to their own families, contribute to their mental burden. Undoubtedly, health care workers are working in a stressful environment that makes them susceptible to burnout syndrome, anxiety, depression, and stress (BADS). Burnout syndrome itself can cause emotional instability, feeling of failure, difficulty in making commitments, and an urge to resign (Maslach et al. 2001).

Several studies reported the psychological impact of the 2003 SARS outbreak among health care workers. The hospital staff experienced the fear of contagion and of spreading the infection to their own family, friends, and co-workers (Maunder et al. 2003, Nickell et al. 2004). Stigmatization and uncertainty were prominent among these individuals (Maunder et al. 2003, Bai et al. 2004). A recent study by Lai et al. (2019) assessing the mental health outcomes of health care workers exposed to COVID-19 patients in Wuhan, China showed that these individuals reported symptoms of anxiety, depression, distress, and insomnia. Notably, these symptoms were adversely severe in nurses and frontline health care workers in comparison to other health care workers. These studies highlight the psychosocial morbidity of disease outbreaks and stress on the need for assessing the psychosocial impact of COVID-19 on health care workers. Furthermore, conducting longitudinal studies are also essential to determine the long-term psychological impact of such outbreaks on health care workers and to identify factors that increase their vulnerability. Such studies will also allow us to assess and develop coping strategies and effective psychosocial support programs to prepare the health care workers for challenges produced by future outbreaks of such nature.

The current study aims to evaluate the mental health outcomes of healthcare workers who are on the frontline of dealing with COVID-19 patients compared to non-COVID-19 patients. We aim to assess the magnitude of symptoms of burnout, depression, anxiety, stress (BADS) and the vulnerability to post-traumatic stress disorder (PTSD) by using established survey-based tools during and after the COVID-19 crisis and performing statistical analysis of the data obtained. The participants include healthcare staff working with COVID-19 patients and those not working with COVID-19 patients as controls, inside and outside Qatar. The study is also expected to be extended internally to assess the psychological impact globally. This study is highly relevant and significant considering previous reports of psychological morbidity of disease outbreaks. It will allow the development of special interventions to provide psychosocial support to the health care workers that would need to be implemented immediately.

ELIGIBILITY:
Inclusion Criteria:

* All healthcare staff working during the COVID-19 outbreak
* Received an email with our electronic survey
* Accepted electronically to participate in our study
* Completed and submitted our electronic questionnaires successfully
* For follow-up: Accepted to receive a follow-up survey

Exclusion Criteria:

* Non-healthcare workers
* Did not accept electronically to participate in our study
* Did not complete not submitted our electronic questionnaires successfully
* For follow-up: Did not accept to receive a follow-up survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to recruit around 25 thousand participants to respond to our online-based survey via email. Participants will include all healthcare staff dealing with COVID-19 patients (group 1), vs. those who are not dealing with COVID-19 patients (group 2), from hospitals and health centers inside and outside Qatar.
  Our questionnaires will be used to assess their mental health by measuring burnout, anxiety, depression and stress levels and post-trauma stress disorder in both groups. Participants' socio-demographic data such as age, gender, profession, marital state, native country, years of experience, weekly working hours will also be collected.
Sampling Method: Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2020-07-11 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
To reflect the effect of COVID-19 on the burnout, anxiety, depression and stress levels of healthcare professionals during the COVID-19 crisis | 6 months
To reflect the effect of COVID-19 on the post-trauma stress disorder levels of healthcare professionals following the COVID-19 crisis | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided